CLINICAL TRIAL: NCT00985452
Title: The Impact of GlowCaps Connect™ and Its Services on Hypertension Medication Adherence: A Randomized Controlled Trial
Brief Title: The Impact of GlowCaps Connect™ and Its Services on Hypertension Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Director, Center for Connected Health, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 2009-P-000254/3;MGH
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Medication Adherence
Keywords: Medication; Adherence; Hypertension
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 2: Intervention (Other): Subjects in Group two will received an activated GlowCaps system, which will remind them to take their medication.
  Interventions: Other: GlowCaps Connect system
- Group 3: Intervention/financial incentive (Other): Subjects in group 3 will receive an activated GlowCaps system, which will provide them with reminders to take their medication, Subjects in group 3 will also receive an additional financial incentive, the amount will be based on how often they remembered to take their medication during the 6-month study.
  Interventions: Other: GlowCaps Connect system
- Group 1: Control (Other): Subjects in group one will receive a de-activated GlowCaps system, which will not provide the reminder service.
  Interventions: Other: Glow cap system - deactivated

INTERVENTIONS:
Other: GlowCaps Connect system — The GlowCaps Connect system is an electronic medication reminder system, which provides reminders to help people to remember to take their medication.
  Other Names: Vitality GlowCaps Connect
  Arms: Group 2: Intervention; Group 3: Intervention/financial incentive
Other: Glow cap system - deactivated — The Glow cap system - deactivated is an electronic medication system, which will track medication adherence.
  Other Names: Vitality GlowCaps
  Arms: Group 1: Control

SUMMARY:
The investigators hypothesize that providing subjects on a once-a-day hypertension medication with GlowCaps ConnectTM will lead to an improvement in their medication adherence. The investigators propose to conduct a 6-month randomized control trial to assess the effect of the GlowCaps Connect™ system on the enhancement of hypertension medication adherence among subjects with a diagnosis of hypertension recruited from the greater Boston area. 130 subjects will be enrolled. Subjects will be randomized into either the control group or into one of two intervention groups.

DETAILED DESCRIPTION:
Participants will use the GlowCap system for 6 months.

Group 1

* The GlowCap bottle provided for subjects in this group will passively track medication adherence over the course of the study
* The pill cap will collect data, but will not provide any visual or auditory alerts
* An Ethernet Gateway connector will collect adherence data from the pill bottle cap via a local wireless network. This data will be sent out of subject's home through the internet.

Group 2

* Subjects in this group will be given daily visual, auditory, and phone call reminders to take their medication via the GlowCap system if they fail to take their hypertension medication at the scheduled dose time
* An Ethernet Gateway connector will collect adherence data from the pill bottle cap via a local wireless network. This data will be sent out of subject's home through the internet.
* Subjects will receive Weekly and Monthly Progress Reports by email and mail, respectively. Reports will include information about medication adherence and target goals. If a subject does not opt-out, Monthly Progress Reports will also be sent to the subject's primary care physician (PCP)
* If the subject chooses, a friend or family member will receive a Weekly Progress Report by email
* If the subject chooses, he/she will receive prompts (via automated telephone call twice a month) to refill his/her prescription
* Subjects demonstrating consistent low adherence to medication will receive additional support in the form of calls from Vitality reminding them to take the medication.

Group 3

* Subjects in this group will be given daily visual, auditory, and phone call reminders to take their medication via the GlowCap system if they fail to take their hypertension medication at the scheduled dose time
* An Ethernet Gateway connector will collect adherence data from the pill bottle cap via a local wireless network. This data will be sent out of subject's home through the internet.
* Subjects will receive Weekly and Monthly Progress Reports by email and mail, respectively. Reports will include information about medication adherence and target goals. If a subject does not opt-out, Monthly Progress Reports will also be sent to the subject's primary care physician (PCP)
* If the subject chooses, a friend or family member will receive a Weekly Progress Report by email
* Subjects will receive financial incentives in the form of a check for meeting a target adherence goal of 80% adherence over each month. The check will be mailed to them at the end of the study.
* If the subjects chooses, he/she will receive prompts (via automated telephone call twice a month) to refill his/her prescription
* Subjects demonstrating consistent low adherence to medication will receive additional support in the form of calls from Vitality reminding them to take the medication and may receive increased financial incentives to meet their target.

Study subjects will attend two study visits, one at the beginning and one at the end of the 6 month period. At these visits they will have their blood pressure recorded and will be asked to complete a survey.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women age 18 and over
* Diagnosis of hypertension
* Take a once a day medication for hypertension
* Internet access via broadband (not dial-up)
* Home router
* A private email account
* Fluency in English (spoken and written)
* Have a Primary Care Physician

Exclusion Criteria:

* People will be excluded if they are not able to adequately respond to researcher's questions or complete the surveys.
* People with significant cognitive deficits will be excluded.
* People will be excluded if they take more than three medications a day for hypertension.
* People will be excluded if they take more than five medications in one day.
* People will be excluded if they have total color blindness.
* People will be excluded if they are both blind and deaf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Quantify the impact of GlowCaps Connect™ and its services on hypertension medication adherence | 6 months

SECONDARY OUTCOMES:
Assess the usability and satisfaction of the GlowCap system | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Kvedar, MD, Principal Investigator — Massachusetts General Hospital